CLINICAL TRIAL: NCT03034551
Title: Randomized Controlled Trial of a Mobile App With Patient Financial Incentives for Tracking and Improving Adherence to Medications & Daily Self-Weighing to Reduce Heart Failure Readmissions
Brief Title: Mobile App With Patient Financial Incentives for Adherence to Heart Failure Medications & Daily Self-Weighing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Wellth Inc. (Industry)
Collaborators: Princeton Healthcare System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: W000002
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Heart Failure; Heart Failure, Congestive; Heart Failure, Systolic
Keywords: Adherence; Financial Incentives; Remote Monitoring; Self-Weighing; Behavioral Economics; Telehealth; mobile health (mHealth); Smartphone App; Wellth App
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Subjects in the treatment arm will be offered a $150 incentive to use the Wellth app each day to log one daily self-weighing and one medication check-in. If a sudden jump in weight is detected among any subjects receiving the Financial Incentive, Mobile Phone App, and Cellular Scale, a UMCPP physician or nurse will then call the patient to assess the patient's symptoms (i.e. increasing shortness of breath or decreases in exertional tolerance, medication and dietary adherence).
  Interventions: Behavioral: Financial Incentive, Mobile Phone App, and Cellular Scale
- Standard of Care (Control) Arm (No Intervention): Patients randomized to the standard of care arm will not receive the Wellth app or scale. They will have the usual discharge instructions as prescribed by their health care team.

INTERVENTIONS:
Behavioral: Financial Incentive, Mobile Phone App, and Cellular Scale — Subjects will be provided a cellular-connected digital scale and will be offered $150 to use the app each day to log one daily self-weighing and one medication check-in. Medication check-ins consist of uploading daily photos of pills at the time of self-administration through the Wellth app. If a 2 lb or greater daily increase in weight, or a 5 lb weekly increase in weight is detected in any patient, a UMCPP physician or nurse will be alerted via automatic email and text. A physician or a nurse will then call the patient to assess the patient's symptoms. If there are increasing heart failure symptoms, the physician or nurse will suggest the patient see their doctor within the next 48 hours and will notify the patient's primary care physician and cardiologist.
  Arms: Intervention Arm

SUMMARY:
The goal of this study is to test the efficacy of a financial incentives-based telehealth intervention to reduce 30- and 90-day heart failure (HF) readmissions by tracking and increasing adherence to patient self-care - specifically by incentivizing adherence to prescribed cardiac medication regimen and daily self-weighing. Patients randomized to the treatment arm will be given a cellular-connected scale to use at home, as well as a mobile app on their smartphone that tracks their adherence to daily self-weighing through the scale and cardiac medications via patient photo submission. The health care team will intervene if a sudden increase in weight is detected (2 lbs/day or 5 lbs/week). Financial incentives of $150 are offered for full adherence over 90 days. Each day where the patient does not step on the scale and complete a medication check-in will result in a deduction of $2 per day from the incentive amount to be paid out. The control group will receive the usual discharge instructions as prescribed by their health care team.

DETAILED DESCRIPTION:
Nonadherence to cardiovascular medications and daily weight monitoring are critical issues in readmissions to the hospital for heart failure. Only 60% of patients adhere to prescribed cardiovascular medications on at least 80% of days, and only 40% monitor their weight daily, despite owning scales. Nationally, nonadherence contributes to excessive HF readmission rates of 50% within 6 months, and 24% within 30 days of discharge. To raise awareness and accountability, the Centers for Medicare & Medicaid Services (CMS) began reporting these rates in 2009, and the Affordable Care Act and value-based contracts with payers have established financial penalties to spur provider-based solutions.

Telehealth interventions are an ideal, low-cost, scalable method to reduce readmissions by remotely enhancing patient support. Telehealth interventions for HF that target medication compliance and self-weighing have demonstrated reductions in readmission rates by 80% or more, but these are not yet widely adopted in clinical practice due to a lack of randomized, controlled studies. We are thus proposing a randomized, controlled study of a proprietary telehealth platform at University Medical Center of Princeton at Plainsboro (UMCPP) to enable remote support for HF patients through a mobile app combined with financial incentives to motivate adherence to medication and self-weighing. Patients admitted to UMCPP with the primary admitting or discharge diagnosis of heart failure with reduced ejection fraction (EF<40%) (ICD-10 codes I50.2_) will be invited to participate in the study.

Each patient in the intervention arm will be offered $150 in incentives along with the Wellth app loaded on to his or her smartphone. When users first log in to the app, which will occur with the guidance of a healthcare provider trained in its use, they will be shown a large dollar amount that they have earned by enrolling in the program - in this study $150 will be offered for 90 days of perfect adherence to medications and daily self-weighing using connected digital scales provided by Wellth. Instructions will also be given stating that missed weight and medication check-ins will result in a $2 deduction per day from the account to be paid out at each monthly pay period.

If a 2 lb. or greater daily increase in weight, or a 5 lb. weekly increase in weight, is detected in any patient, a UMCPP physician or nurse will be alerted via automatic email and text. A physician or a nurse will then call the patient to assess the patient's symptoms (i.e. increasing shortness of breath or decreases in exertional tolerance, medication and dietary adherence). Once a weight gain alert has been triggered, the team will continue to receive additional data about the patient for the next 7 days to see if weight continues to increase which would trigger an additional phone call and patient physician notification.

After a call is made to the patient, if, in the clinical judgment of the physician or nurse that there are increasing heart failure symptoms, the physician or nurse will suggest to the patient that they make an appointment and see their doctor within the next 48 hours.

Benefits of this study to the intervention arm include better health, reduced risk of readmission, and concomitant reduction in healthcare burden, as well as a small but tangible financial gain. Benefits for society, assuming widely applicable success, include reduction in population-wide readmission rates due to greater health, and reduction in healthcare spending.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to or discharged from University Medical Center of Princeton at Plainsboro (UMPCC) with the primary diagnosis of heart failure with reduced ejection fraction (ICD-10 code I50.2x)
* Standard of care medications for heart failure with reduced ejection fraction
* Own a smart phone with a sufficient data plan or home Wi-Fi. Up to 30 phones can be provided if needed.
* Able to speak and understand either English or Spanish and able to learn the Wellth app.

Exclusion Criteria:

* Diagnosis of HF following non-cardiac admission
* Discharge to a care facility (anywhere that is not home)
* Inability to step on a scale and steady oneself to obtain an accurate weight
* Cognitive impairment or documented psychiatric illness that limits ability to understand and respond to health-related questions
* Inability to operate a mobile phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
30-Day Cardiac Readmissions | 30 Days
  Average rates of hospital readmissions within 30 days assessed by medical record review and patient interviews

SECONDARY OUTCOMES:
90-Day Cardiac Readmissions | 90 Days
  Average rates of hospital readmissions within 90 days assessed by medical record review and patient interviews
Adherence to Daily Medications | 90 Days
  The percentage of days for which a patient submitted medication photos in the 90 days following discharge
Adherence to Daily Self-Weighings | 90 Days
  The percentage of days for which a patient completed a self-weighing using the provided cellular-connected scale in the 90 days following discharge

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Bergmann, MD, PhD, Principal Investigator — Princeton Healthcare System
Locations (1):
- University Medical Center of Princeton at Plainsboro, Plainsboro, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ho PM, Bryson CL, Rumsfeld JS. Medication adherence: its importance in cardiovascular outcomes. Circulation. 2009 Jun 16;119(23):3028-35. doi: 10.1161/CIRCULATIONAHA.108.768986. PMID 19528344
- [Background] van der Wal MH, Jaarsma T, Moser DK, Veeger NJ, van Gilst WH, van Veldhuisen DJ. Compliance in heart failure patients: the importance of knowledge and beliefs. Eur Heart J. 2006 Feb;27(4):434-40. doi: 10.1093/eurheartj/ehi603. Epub 2005 Oct 17. PMID 16230302
- [Background] Desai AS, Stevenson LW. Rehospitalization for heart failure: predict or prevent? Circulation. 2012 Jul 24;126(4):501-6. doi: 10.1161/CIRCULATIONAHA.112.125435. No abstract available. PMID 22825412
- [Background] Maric B, Kaan A, Ignaszewski A, Lear SA. A systematic review of telemonitoring technologies in heart failure. Eur J Heart Fail. 2009 May;11(5):506-17. doi: 10.1093/eurjhf/hfp036. Epub 2009 Mar 29. PMID 19332417
- [Background] Maeng DD, Starr AE, Tomcavage JF, Sciandra J, Salek D, Griffith D. Can telemonitoring reduce hospitalization and cost of care? A health plan's experience in managing patients with heart failure. Popul Health Manag. 2014 Dec;17(6):340-4. doi: 10.1089/pop.2013.0107. PMID 24865986
- [Background] Haff N, Patel MS, Lim R, Zhu J, Troxel AB, Asch DA, Volpp KG. The role of behavioral economic incentive design and demographic characteristics in financial incentive-based approaches to changing health behaviors: a meta-analysis. Am J Health Promot. 2015 May-Jun;29(5):314-23. doi: 10.4278/ajhp.140714-LIT-333. PMID 25928816
- [Background] Chaudhry SI, Wang Y, Concato J, Gill TM, Krumholz HM. Patterns of weight change preceding hospitalization for heart failure. Circulation. 2007 Oct 2;116(14):1549-54. doi: 10.1161/CIRCULATIONAHA.107.690768. Epub 2007 Sep 10. PMID 17846286